CLINICAL TRIAL: NCT06799390
Title: Vagus Nerve Stimulation Following Intracerebral Hemorrhage (IHC) to Mitigate ICH-induced Inflammation and Cerebral Edema
Brief Title: Auricular VNS Following Intracerebral Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202408166
Record Dates: First submitted 2025-01-13; First posted 2025-01-29 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Intracerebral Hemorrhage
Keywords: vagal nerve stimulation; pathologic processes; intracerebral hemmorrhage; cerebrovascular disorders; brain diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage; Pathologic Processes; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either stimulation or sham stimulation arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants will be fitted with an auricular stimulator, but blinded to whether they are receiving stimulation or not. Outcome scores will be assessed and recorded by clinicians blinded to treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Auricular VNS Stimulation (Experimental): Participants receive twice daily auricular vagal nerve stimulation
  Interventions: Device: Auricular Vagus Nerve Stimulation
- Sham Auricular VNS Stimulation (Sham Comparator): Participants will have an auricular vagal nerve stimulator placed in their ear twice daily, without the stimulation applied
  Interventions: Device: Sham Auricular Vagus nerve Stimulation

INTERVENTIONS:
Device: Auricular Vagus Nerve Stimulation — Transcutaneous auricular vagal nerve stimulation
  Arms: Auricular VNS Stimulation
Device: Sham Auricular Vagus nerve Stimulation — Transcutaneous auricular vagal nerve ear clip applied without current
  Arms: Sham Auricular VNS Stimulation

SUMMARY:
This study will evaluate whether non-invasive auricular vagal nerve stimulation lowers inflammatory markers, and improves outcomes following intracerebral hemorrhage.

DETAILED DESCRIPTION:
Vagal nerve stimulation (VNS) has been studied as a novel method of reducing inflammation, and it has been successfully used in animal models of inflammatory conditions. The purpose of the proposed study is to determine if transcutaneous auricular VNS will impact inflammatory markers in the blood and cerebrospinal fluid (CSF) in patients with intracerebral hemorrhage, and how it impacts their clinical course and outcomes.

This study will involve randomizing patients to stimulation with VNS, or sham stimulation. Blood and CSF will be collected on admission, and serially throughout the patient's admission. Clinical events tracked during the hospital stay include the development of peri-hematomal edema, interventions for edema (medical or surgical), and intensive care unit and hospital stay. Outcomes following admission will include functional scores at discharge, and at follow-up visits for up to 2 years after discharge. No additional appointments will be made specially for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who present with a spontaneous supratentorial intracerebral hemorrhage (ICH) to Barnes Jewish Hospital

Exclusion Criteria:

* Patients < 18 years old
* Patients with a presumed traumatic etiology for their ICH, infratentorial location, ICH volume > 60 ml or < 10 ml, at risk of imminent death (e.g. Glasgow Coma Scale, GCS of 3 or one or more pupils unreactive), surgical intervention imminently planned (not including ventriculostomy)
* Patients undergoing active cancer therapy
* Patients with sustained bradycardia on arrival with a heart rate < 50 beats per minute.
* Patients who cannot be enrolled within 48 hours of the initial bleed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2030-02-09 (Estimated); Study Completion 2032-02-09 (Estimated)

PRIMARY OUTCOMES:
Change in the inflammatory marker IL-6 in plasma | 14 days
  Blood samples collected on days 1, 4, 7, 10, and 14 (Day 1 serves as baseline, prior to first treatment). Inflammatory markers will be reported in pg/mL.
Growth of perihematomal edema | 14 days
  Change in edema extension distance (baseline vs. peak) will be compared between groups, via quantitative assessment of serial computed tomography (CT) scans obtained on day 1, 4, 7, 10, and 14 (Day 1 serves as baseline, prior to first treatment).
Neurological worsening | Through hospital admission, average 14 days
  Occurrence of clinical deterioration due to edema by criteria of 1) a reduction in GCS by 2 points or greater that persists for at least one hour, 2) worsening focal neurological deficits (NIHSS increase by at least 4 points), excluding other causes, or 3) need for surgical intervention or medical treatments for edema (osmotic therapies).

SECONDARY OUTCOMES:
Change in additional inflammatory markers in plasma | 14 days
  Blood samples collected on days 1, 4, 7, 10, and 14 to evaluate for IL-1b, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-17a, GM-CSF, IFN gamma, and TNF-α. Inflammatory markers will be reported in pg/mL.
Change in inflammatory markers in cerebrospinal fluid | 14 days
  Cerebrospinal fluid samples collected on days 1, 4, 7, 10, and 14 to evaluate for IL-1b, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-17a, GM-CSF, IFN gamma, and TNF-α. Inflammatory markers will be reported in pg/mL.
Relative perihematomal edema | 14 days
  Relative perihematomal edema volume, the ratio of perihematoma volume to intracerebral hematoma volume
Neurological outcome | 2 years
  Modified Rankin Scale for Neurological Disability (minimum score 0, maximum score 6, better outcomes have lower scores)
Hospital length of stay | Through hospital admission, average 14 days
  Total length of stay in the hospital, and in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Eric Leuthardt, MD MBA, Study Chair — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huguenard AL, Tan G, Rivet DJ, Gao F, Johnson GW, Adamek M, Coxon AT, Kummer TT, Osbun JW, Vellimana AK, Limbrick DD, Zipfel GJ, Brunner P, Leuthardt EC. Auricular Vagus Nerve Stimulation Mitigates Inflammation and Vasospasm in Subarachnoid Hemorrhage: A Randomized Trial. medRxiv [Preprint]. 2024 May 1:2024.04.29.24306598. doi: 10.1101/2024.04.29.24306598. PMID 38746275
- [Background] Huguenard A, Tan G, Johnson G, Adamek M, Coxon A, Kummer T, Osbun J, Vellimana A, Limbrick D Jr, Zipfel G, Brunner P, Leuthardt E. Non-invasive Auricular Vagus nerve stimulation for Subarachnoid Hemorrhage (NAVSaH): Protocol for a prospective, triple-blinded, randomized controlled trial. PLoS One. 2024 Aug 23;19(8):e0301154. doi: 10.1371/journal.pone.0301154. eCollection 2024. PMID 39178291
- [Background] Tan G, Huguenard AL, Donovan KM, Demarest P, Liu X, Li Z, Adamek M, Lavine K, Vellimana AK, Kummer TT, Osbun JW, Zipfel GJ, Brunner P, Leuthardt EC. The effect of transcutaneous auricular vagus nerve stimulation on cardiovascular function in subarachnoid hemorrhage patients: A randomized trial. Elife. 2025 Jan 9;13:RP100088. doi: 10.7554/eLife.100088. PMID 39786346